CLINICAL TRIAL: NCT05180136
Title: Efficacy and Tolerability of Rice Bran Extract in Mildly to Moderately Depressed Patients: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Efficacy of Rice Bran Extract in Mildly to Moderately Depressed Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2021-031
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rice bran extract group (Experimental): This group takes rice bran extract for 8 weeks.
  Interventions: Dietary Supplement: Rice bran extract group
- Control group (Placebo Comparator): This group takes a placebo for 8 weeks.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Rice bran extract group — Rice bran extract 1,000 mg/day for 8 weeks
  Arms: Rice bran extract group
Dietary Supplement: Control group — Placebo 1,000 mg/day for 8 weeks
  Arms: Control group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects and tolerability of rice bran extract on depressive symptoms and related biomarkers in mildly to moderately depressed patients for 8 weeks.

DETAILED DESCRIPTION:
A previous animal study has indicated that rice bran extract provided inhibition of MAO-B enzyme activity and ROS formation in a corticosterone-induced depression-like animal model. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of rice bran extract on depressive symptoms and related biomarkers in mildly to moderately depressed patients for 8 weeks; the safety of the compound is also evaluated. The Investigators examine the Korean version of the Hamilton Depression Rating Scale, the Korean Version of the Beck-II Depression Inventory, the Korean version of the Patient Health Questionnaire-9, the Perceived Stress Scale, the Korean version of the Beck Anxiety Inventory and biomarkers at baseline and after 8 weeks of intervention. One hundred adults were administered either 1,000 mg of rice bran extract or a placebo each day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

- the Korean version of the Hamilton Depression Rating Scale score between 7-24

Exclusion Criteria:

* No depressive symptom (K-HRSD ≤ 6) or severely depressed (K-HRSD ≥ 25)
* Those are taking hormone therapy such as estrogen within the past 6 months
* Those are taking the following drugs within the last 1 month or need to take them during the study period (sleep aids, antidepressants, selective estrogen receptor modulators, etc.)
* Those with a history of treatment for depression
* Abnormal liver or renal function (more than twice the normal upper limit of the research institute)
* Uncontrolled diabetes mellitus (>160 mg/dL of fasting blood sugar)
* Uncontrolled hypertension (>160/100 mmHg)
* Uncontrolled thyroid diseases.
* Those who are taking drugs, functional foods, herbs, etc. that may affect depression
* Alcohol abuser
* Allergic reaction to this test food
* Those who participated in other drug clinical trials within 1 month from the screening date.
* Severe gastrointestinal symptoms such as heartburn and indigestion
* Those who are pregnant, lactating, or plan to become pregnant during the clinical trial
* Those who are judged to be unsuitable by the PI for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The Korean version of the Hamilton Depression Rating Scale (K-HDRS) | 8 weeks
  using K-HDRS score. The minimum score was 0 and the maximum score was 50, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The Korean Version of the Beck-II Depression Inventory (K-BDI II) | 8 weeks
  using K-BDI II score. The minimum score was 0 and the maximum score was 63, and higher scores mean a worse outcome.
The Korean version of the Patient Health Questionnaire-9 (K-PHQ-9) | 8 weeks
  using K-PHQ-9 score. The minimum score was 0 and the maximum score was 27, and higher scores mean a worse outcome.
The Korean version of the Beck Anxiety Inventory (K-BAI) | 8 weeks
  using K-BAI score. The minimum score was 0 and the maximum score was 63, and higher scores mean a worse outcome.
The Korean of the Perceived Stress Scale(K-PSS) | 8 weeks
  using K-PSS score. The minimum score was 0 and the maximum score was 40, and higher scores mean a worse outcome.
serotonin concentration (nM) | 8 weeks
  Change during 8 weeks
Brain-derived neurotrophic factor concentration (ng/ml) | 8 weeks
  Change during 8 weeks
salivary cortisol concentration (U/mL) | 8 weeks
  Change during 8 weeks
dopamine concentration (pg/μL) | 8 weeks
  Change during 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh SY, Lee YL, Kim SH, Lee SY. Efficacy of rice bran extract for alleviating depressive symptoms in adults: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2025 Jul;122(1):112-121. doi: 10.1016/j.ajcnut.2025.05.021. Epub 2025 May 21. PMID 40409466